CLINICAL TRIAL: NCT01563263
Title: A Confirmatory Phase II/III Study Assessing Efficacy, Immunogenicity and Safety of IC43 Recombinant Pseudomonas Vaccine Intensive Care Patients
Brief Title: Confirmatory Phase II/III Study Assessing Efficacy, Immunogenicity and Safety of IC43
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC43-202
Record Dates: First submitted 2012-03-14; First posted 2012-03-26 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Pseudomonas Aeruginosa Infection
Keywords: IC43; Pseudomonas Aeruginosa; mechanically ventilated ICU patients; ICU patients
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IC43 100 mcg (Active Comparator): IC43 100 mcg intramuscular injection, IC43 is a recombinant Pseudomonas aeruginosa fusion protein
  Interventions: Biological: IC43
- Placebo (Placebo Comparator): phosphate buffered saline solution containing 0,9 % NaCL
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: IC43 — 100 mcg
  Other Names: Pseudomonas Aeruginosa
  Arms: IC43 100 mcg
Drug: Placebo — phosphate buffered saline (PBS) solution containing 0,9 % NaCl
  Other Names: phosphate buffered saline (PBS)
  Arms: Placebo

SUMMARY:
This is a confirmatory, randomized, placebo-controlled, multi-center, double-blinded phase II/III study. The study population consists of male or female intensive care unit (ICU) patients with a need for mechanical ventilation for more than 48 hours, aged between 18 and 80 years.

DETAILED DESCRIPTION:
This is a confirmatory, randomized, placebo-controlled, multi-center, double-blinded phase II/III study. The study population consists of male or female intensive care unit (ICU) patients with a need for mechanical ventilation for more than 48 hours, aged between 18 and 80 years.

Eight-hundred patients will be enrolled at approximately 50 study centers. Informed consent (i.e., from the patient or from the patient's legally authorized representative) or waiver will be obtained according to regional requirements prior to any study related procedures. Patients will be randomized to receive either IC43 100 mcg or placebo and will receive the first vaccination on Day 0. The second vaccination will be applied on Day 7. In case ICU discharge occurs before Day 7, immunization will be done at the hospital ward.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients admitted to an intensive care unit (ICU) with need for mechanical ventilation for at least 48 hours, aged between 18 and 80 years at Visit 0
* written informed consent or waiver according to the national regulations
* no childbearing potential or negative pregnancy test

Exclusion Criteria:

* Sequential Organ Failure Assessment (SOFA) < 4 on Day 0
* Patients <6 months post organ transplantation
* readmission to ICU during the current total hospital stay on Day 0
* patients admitted to ICU within 2 days after surgery
* patients admitted to ICU due to trauma
* elective surgery until Day 28 after first vaccination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
number of deaths until Day 28 | until Day 28

SECONDARY OUTCOMES:
number of deaths in comparison on Day 14, 56 and 90 | until Day 90
number of deaths onDay 28, 56 and 90 in patients surviving Day 14 and receiving IC43 or placebo | until Day 90
number of deaths on Day 14, 28, 56 and 90 in patients surviving Day 3 and receiving IC43 or placebo | until Day 90
number of overall survival in all patients and in patients surviving Day 14 | until Day 180
number of deaths related to sepsis at Day 14, 28, 56 and 90 in patients receiving IC43 or placebo | until Day 90
number of surviving subjects after Sepsis receiving IC43 or placebo | until Day 180
number of deaths in patients in-ICU and in-hospital receiving IC43 or placebo until Day 14, 28, 56,90, 180 | until Day 180
percentage of patients with invasive infection with P. aeruginosa, such as bacteremia or P. aeruginosa urinary tract infection in patients receiving IC43 or placebo up to Day 56 after first vaccination | until Day 56
percentage of patients with P. aeruginosa respiratory tract infection or P. aeruginosa respiratory tract colonization in patients receiving IC43 or placebo up to Day 56 after first vaccination | until Day 56
Organ function in patients receiving IC43 or placebo during ICU stay | during ICU stay
Days of ICU stay in patients receiving IC43 or placebo | Until Day 180
Immunogenicity at Day 7, 14, 28, 56 and 180 as determined by OprF/I specific IgG antibody titer measured by ELISA in patients receiving IC43 or placebo | until Day 180
Number of SAEs and AEs during the vaccination period up to 180 days after the first vaccination | until Day 180
systemic tolerability | until Day 7
  blood pressure
number of local reactions at the injection site | until Day 180
Composite measure of laboratory parameters | until Day 56
systemic tolerability | until Day 7
  pulse
systemic tolerability | until Day 7
  body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eder, Mag, Study Chair — Valneva Austria GmbH
Locations (50):
- Austria (6):
  - LKH - University Clinic Graz, Graz, Graz
  - LKH Salzburg, Salzburg, Salzburg
  - Medical University of Vienna, Vienna, Vienna
  - Otto Wagner Spital, Vienna, Vienna
  - Wilhelminenspital & Kaiserin-Elisabeth-Spital, Vienna, Vienna
  - Krankenhaus Hietzing, Vienna
- Belgium (6):
  - ULB Hospital Erasme, Brussels, Brussels Capital
  - University Hospital Brussels, Brussels, Brussels Capital
  - Hospital Saint Luc, Brussels, Brussels Capital
  - Ziekenhuis Oost Limburg, Genk, Genk
  - University Hospital Ghent, Ghent, Ghent
  - Clinique St. Pierre, Ottignies, Ottignies
- Czechia (7):
  - Faculty Hospital St. Ann, Brno, Brno
  - Faculty Hospital, Hradec Krakove, Hradec Krakove
  - Faculty Hospital Kralovske Vinohrady, Prague, Prague
  - Faculty Hospital Motol, Prague, Prague
  - Central Military Hospital, Prague, Prague
  - Fakultní nemocnice Olomouc, Olomouc
  - Krajská nemocnice T. Bati, a.s., Zlín
- Germany (14):
  - HELIOS Klinikum Aue, Aue, Aue
  - Carl-Thiem-Klinikum Cottbus, Cottbus, Cottbus
  - Städtisches Klinikum Dessau, Dessau, Dessau-Roßlau
  - Klinikum Dortmund, Dortmund, Dortmund
  - Neurologische Universitätsklinik, Dresden, Dresden
  - HELIOS Klinikum Erfurt, Erfurt, Erfurt
  - Helios Kreikrankenhaus Gotha/Ohrdruf, Gotha, Gotha
  - Bermannstrost BG Kliniken Halle, Halle, Halle/Saale
  - Saarland University Hospital, Homburg/Saar, Homburg/Saar
  - Universitätsklinikum Schleswig-Holstein, Kiel, Kiel
  - Klinikum rechts der Isar, München, München
  - HELIOS Klinikum Berlin-Buch, Berlin, State of Berlin
  - Charite-Universitätsmedizin Berlin, Berlin, State of Berlin
  - HELIOS Klinikum Wuppertal, Wuppertal, Wuppertal
- Hungary (10):
  - St. Imre Hospital, Budapest, Budapest
  - Uzsoki Hospital, Budapest, Budapest
  - Kenezy Korhaz Debrecen, Debrecen, Debrecen
  - Debreceni Egyetem OEC Kazincbarcikai Korhaz, Kazincbarcika, Kazincbarcika
  - Flor Ferenc Korhaz Hospital, Kistarcsa, Kistarcsa
  - University of Pecs, Pécs, Pecs
  - University of Szeged, Szeged, Szeged
  - Fejer County Hospital, Székesfehérvár, Szekesfehervar
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Pécsi Tudományegyetem Neurológiai Klinika, Pécs
- Spain (7):
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario de Getafe, Madrid, Madrid
  - University Hospital Marques de Valdecilla, Santander Cantabria, Santander Cantabria
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Universitario y Policlínico La Fe, Valencia

REFERENCES:
- [Derived] Adlbrecht C, Wurm R, Depuydt P, Spapen H, Lorente JA, Staudinger T, Creteur J, Zauner C, Meier-Hellmann A, Eller P, Laenen MV, Molnar Z, Varkonyi I, Schaaf B, Hejja M, Sramek V, Schneider H, Kanesa-Thasan N, Eder-Lingelbach S, Klingler A, Dubischar K, Wressnigg N, Rello J. Efficacy, immunogenicity, and safety of IC43 recombinant Pseudomonas aeruginosa vaccine in mechanically ventilated intensive care patients-a randomized clinical trial. Crit Care. 2020 Mar 4;24(1):74. doi: 10.1186/s13054-020-2792-z. PMID 32131866